CLINICAL TRIAL: NCT05775393
Title: Effects of Adding Dexamethasone Plus Ketamine to Bupivacaine for Ultrasound Guided Serratus Plane Block as Analgesia in Major Breast Surgery
Brief Title: Effects of Adding Dexamethasone Plus Ketamine to Bupivacine in Serrtatus Plane Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Fakher Mohamed Abdou, Dr, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AP2202-30105
Record Dates: First submitted 2023-02-21; First posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Pain
Keywords: Serratus ,analgesia ,ketamine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Serratus anterior plane block using 30ml of (bupivacaine 0 .25 % and dexamethasone 4 mg)
  Interventions: Procedure: Serratus anterior plane block for MRM
- Group B (Experimental): Serratus anterior plane block using 30ml of (bupivacaine 0.25% and dexamethasone 4mg with ketamine 50 mg).
  Interventions: Procedure: Serratus anterior plane block for MRM

INTERVENTIONS:
Procedure: Serratus anterior plane block for MRM — They will randomly assigned to two groups of 30 patients each, at 1:1 allocation ratio using computer-generated random numbers concealed in sealed opaque envelopes.
  Group (A):
  Patients will receive ultrasound-guided serratus anterior block using 30ml of (bupivacaine 0 .25 % and dexamethasone 4 mg).
  Group (B):
  Patients will receive ultrasound-guided serratus anterior block using 30ml of (bupivacaine 0.25% and dexamethasone 4mg with ketamine 50 mg).
  All the medications were prepared by an anesthesiologist not participating in the study.

SUMMARY:
This randomized, double-blind trial included 60 female patients undergoing modified radical mastectomy. The study carried out at National Cancer Institute, cairo university after approval of the local ethical committee.

The study aiming to compare the analgesic efficiency of adding dexamethasone or ketamine plus dexamethasone to bupivacaine in ultrasound-guided serratus anterior plane block (SAPB) performed with modified radical mastectomy surgery.

DETAILED DESCRIPTION:
They will randomly assigned to two groups of 30 patients each, at 1:1 allocation ratio using computer-generated random numbers concealed in sealed opaque envelopes.

Group (A):

Patients will receive ultrasound-guided serratus anterior block using 30ml of (bupivacaine 0 .25 % and dexamethasone 4 mg).

Group (B):

Patients will receive ultrasound-guided serratus anterior block using 30ml of (bupivacaine 0.25% and dexamethasone 4mg with ketamine 50 mg).

All the medications were prepared by an anesthesiologist not participating in the study.

Preoperative visit :

All cases will be assessed for any hemodynamic abnormalities in the preoperative room. Patient will be informed about the purpose and the content of the study before surgery. An informed consent |will be obtained from the participants.

Anesthetic technique :

General anesthesia A uniform anesthetic technique was used in two groups, namely, after pre oxygenation with 100% oxygen for 3 mints, induction of anesthesia will be by IV propofol 2 mg/kg, fentanyl 200 μg and atracurium 0.5 mg/kg to facilitate endotracheal intubation.

Anesthesia will be maintained with isoflurane 1-2% in 50% air in oxygen mixtures. Intermittent dose of atracurium for muscle relaxation and fentanyl will be used if heart rate increased more than 20% of initial HR.

All patients will be mechanically ventilated to maintain end-tidal carbon dioxide tension around 35 mmHg.

After induction of general anesthesia, ultrasound-guided SAPB will be done. Technique of SAPB Patients will be placed in the lateral position with the diseased side up. A linear ultrasound transducer (10-12 MHz) is placed over the mid-clavicular region of the thoracic cage in a sagittal plane.

The fifth rib is identified in the mid-axillary line. The following muscles are identified easily overlying the fifth rib: the latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscle (deep and inferior).

As an extra-reference point, the thoracodorsal artery is used to aid the identification of the plane superficial to the serratus muscle.

The needle (22G, 50-mm Tuohy needle) is introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus muscle.

Under continuous ultrasound guidance, local anesthetic solution is injected and fanning of local anesthetic is observed.

All patients will be continuously monitored with 5 leads electrocardiogram (ECG), pulse oximetry, non-invasive blood pressure monitoring (NIBP), end-tidal CO2, and TOF.

Inhalation anesthetic will be discontinued at the end of surgery and neuromuscular blockade was reversed by IV injection of neostigmine 0.05 mg/kg with atropine 0.01 mg/kg after fulfilling the criteria for extubation. Patients were extubated and transferred to surgical ICU.

For postoperative pain management, all patients will receive intravenous (IV) paracetamol 1 gm every 6 hrs (Injectemol, Pharco B International, Pharma-tech) then morphine IV (2-4 mg) if required to keep VAS score less than 3.

Morphine consumption during the first 24 postoperative hours as a rescue drug was calculated.

Patients will be continuously monitored for heart rate, oxygen saturation and systemic blood pressure and we will record every 10 min for the initial 1 hr. of the blockade; every 30 mints for the next 2 hrs. And then 2 hourly for the next 12 hrs.

As soon as the patient is alert enough, VAS score of pain (10 mm vertical scale from 0 to 10 where zero means no pain and 10 is the worst pain) was recorded every 2 hrs.

Sedation was assessed using the observer's assessment of alertness/sedation (OAA/S) scale.

The scale was scored as a composite score ranging from 1 (deep sleep) to 5 (alert).

Signs of morphine side effects (nausea, vomiting, dizziness, an unusual pleasant feeling, sweating, headache, anxiety, and constipation) will be monitored.

In case of nausea and/or vomiting, 10 mg metoclopramide was given intravenously.

Signs of side effects of SAPB as dyspnea, chest pain in case of pneumothorax and signs of local anesthetic toxicity will be monitored as arrhythmias , convulsions and circulatory collapse

ELIGIBILITY:
Inclusion Criteria:

* All female patient undergoing modified radical mastectomy
* Age from 20 to 60 years
* ASA physical status I,II and III class

Exclusion Criteria:

* Refusal for SAPB.
* Defective coagulation.
* Infection at the site of injection.
* History of allergy to the study drugs

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Post ooerative analgesia requirment | 24 hours
  Total post-operative morphine consumption over the first 24 hours post-operative and difference between two groups.
Time of first analgesic request | 24 hours
  The time to first request of analgesic postoperatively and difference between two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Fakher, Cairo, Matareya, Egypt